CLINICAL TRIAL: NCT03822455
Title: A Phase 2b Randomised, Double-blind, Parallel-group Study of Alginate Oligosaccharide (OligoG) Dry Powder Inhalation in Addition to Standard of Care Compared to Placebo in Addition to Standard of Care in Patients with Cystic Fibrosis (CF)
Brief Title: A Phase 2b Randomised, Placebo Controlled Study of OligoG in Patients with Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: AlgiPharma AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORDCF205
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Randomised, double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomised to receive OligoG or placebo DPI. The investigational medicinal products will have identical appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OligoG DPI (Active Comparator): Active DPI containing the oligosaccharide OligoG and excipients
  Interventions: Drug: OligoG DPI
- Placebo DPI (Placebo Comparator): Placebo DPI containing lactose and excipients
  Interventions: Drug: OligoG DPI

INTERVENTIONS:
Drug: OligoG DPI — OligoG Dry Powder for Inhalation

SUMMARY:
A double-blind, randomised study of OligoG DPI compared to placebo DPI, both on top of standard-of-care, to assess safety, efficacy and tolerability. Adult patients with Cystic Fibrosis will be included in the study.

DETAILED DESCRIPTION:
The alginate oligosaccharide OligoG CF-5/20 dry powder for inhalation (OligoG DPI) represents a novel therapeutic approach for patients with cystic fibrosis (CF). OligoG has been shown to release stagnant mucus, modulate sputum rheology and disrupt the biofilm formation often typically observed in CF. These properties will in turn facilitate mucus clearance and promote effectiveness of antibiotic therapy against the chronic pulmonary infections characteristic of CF.

Patients with CF (age 18 years or older) will be eligible to participate in this study.

The design will be a randomised, blinded, placebo-controlled pilot study for proof of concept that OligoG DPI can improve lung function in adult CF patients. Study medication will be given twice daily for twelve weeks on top of standard of care (SOC). Thirty-three patients will be included, out of which twenty-two shall receive OligoG, and eleven shall receive placebo.

After all patients have completed the 12 week double blind treatment period, all patients will be offered open-label OligoG twice daily, in addition to standard of care, for 12 months.

The primary endpoint will be absolute change i percent predicted FEV1

Exploratory parameters will include sputum microbiology.

ELIGIBILITY:
Inclusion Criteria:

* Genotypic confirmation of CFTR mutation or clinical diagnosis of Cystic Fibrosis (CF) confirmed by a sweat chloride value ≥60 mmol/L by quantitative pilocarpine iontophoresis.
* Age 18 years or older.
* Male or female patients with any ethnicity.
* FEV1 at screening in the range of ≥40% and 90% of the predicted normal for age, sex, and height, according to the GLI equation (Eur Respir J. Dec 2012; 40(6): 1324-1343).
* History of Pseudomonas aeruginosa (PA) infection with at least one positive microbiological PA testing during the last 12 months before the Screening Visit.
* History of antibiotic treatment due to PA infection (not for eradication therapy) during the last 12 months
* Concomitant treatment with inhaled tobramycin, colistin, or aztreonam (either cycled or continuous) for at least 3 months at screening to treat PA infection. In case of cycled antibiotic treatment, the treatment should start with an active cycle at the day of randomisation (+/- 2 day) (together with the IMP intake). If taking tobramycin cycled with another antibiotic, IMP should start on the active cycle of tobramycin.
* Stable CF disease as judged by the investigator.
* Willing to remain on a stable CF medication regimen (standard of care; SOC) during the study.
* Women of child-bearing potential must have a negative urine pregnancy test at the Screening and Randomisation Visit.
* Male and female patients must use acceptable contraceptive methods for the duration of the study. Male and female patients without child-bearing potential (i.e. who are infertile, surgically sterile or post-menopausal) are exempted from the contraceptive requirements. For the purpose of this study acceptable contraception is defined as one or a combination of the following:

  * oral, injected, transdermal or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Capable of inhaling dry powder.
* Willing to sign informed consent
* Willing and able to follow the study procedures.

Exclusion Criteria:

* Use of hypertonic saline more than 2 times a day. If hypertonic saline is used, OligoG inhalation should be taken at least 15 minutes after completion of hypertonic saline therapy.
* Use of CFTR modulator therapies.
* Clinically significant abnormal findings of haematology or clinical chemistry;

  * Elevated gamma GT (GGT), ALT, or AST > 3x the upper normal limit of normal (ULN)
  * Bilirubin >2x ULN
  * Abnormal renal function, with a creatinine clearance calculated <50ml/min
  * Haemoglobin <10g/dL
* History of any comorbidity that, in the opinion of the investigator, might distort the results of the study or cause an additional risk in administering study drug to the patient.
* Pulmonary exacerbation within 28 days prior to randomisation.
* Change in CF therapy within 28 days before randomisation (first dose of IMP).
* Pregnant or breastfeeding females.
* History of allergic reactions to the ingredients of the IMP according to Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or 4, including lactose and milk protein.
* Patients unable to perform pulmonary function tests according to the ATS/ERS criteria.
* Uncontrolled or unstable chronic diseases (e.g. congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations) that would limit the compliance with study requirements in the opinion of the investigator.
* Any acute illness in the last 14 days
* History of, or planned organ transplantation.
* Lung infection with organisms associated with a more rapid decline in pulmonary status (including, but not limited to Burkholderia cenocepacia, Burkholderia dolosa, and Mycobacterium abscessus). For subjects who have had a history of a positive culture, the following criteria will be used to determine whether the subject is free of infection with such organisms:-

  * The subject has not had a respiratory tract culture positive for these organisms within the 12 months before the date of informed consent, and
  * The subject has had at least 2 respiratory tract cultures negative for such organisms within the 12 months before the date of informed consent, with the first and last of these separated by at least 3 months, and the most recent one within the 6 months before the date of informed consent.
* Active allergic bronchopulmonary aspergillosis (ABPA) in the last 12 months prior to the Screening Visit, that has received pharmacological treatment for ABPA.
* Requirement for continuous (24 hour/day) oxygen supplementation.
* Patients currently receiving any other investigational treatment, or who have participated in a clinical study within 4 weeks (28 days) prior to the screening visit.
* Current malignant disease (with the exception of basal cell carcinoma and cervical neoplasia).
* Any medical or psychological condition, other than CF, which in the opinion of the investigator exposes the patient to an unacceptably high risk.
* Patients with documented or suspected, clinically significant, alcohol or drug abuse as per Investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
FEV1 percent predicted | Baseline compared to 12 weeks
  Absolute change in percent Forced Expiratory Volume in one second,

SECONDARY OUTCOMES:
Pulmonary exacerbation rate | 6 months before treatment, 6 months after treatment,
  rate of pulmonary exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wark, Principal Investigator — John Hunter Hospital
Locations (1):
- John Hunter Hospital, Newcastle, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No